CLINICAL TRIAL: NCT00021580
Title: Modification of the "Edmonton Protocol" to Allow for Successful Islet Transplantation From a Single Pancreas and Extension of the "Edmonton Protocol" to Kidney Transplant Recipients (Project 1 of JDFI Washington University Center for Islet Transplantation)
Brief Title: Modification of the "Edmonton Protocol" to Allow for Successful Islet Transplantation From a Single Pancreas and Extension of the "Edmonton Protocol" to Kidney Transplant Recipients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00036-0775
Record Dates: First submitted 2001-07-24; First posted 2001-07-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Procedure: human cadaveric islet cell transplantation

SUMMARY:
The experience of the Edmonton Group with islet transplantation and use of the "Edmonton Protocol" provides much promise for T1DM patients. However, the need to use 2 or more donor pancreases to achieve freedom from insulin shots limits the widespread use of this protocol. Two classes of oral antidiabetic drugs improve insulin action and reduce the amount of insulin needed to have normal blood sugars. The first part of the proposed project (Group 1) will use these drugs in conjunction with the Edmonton Protocol to allow for successful islet transplantation from islets isolated from a single pancreas.

The Edmonton Protocol is a treatment, not a cure. It requires the long-term use of powerful immunosuppressive drugs that are expensive and increase the risk of infection and cancer. T1DM patients who have a functioning kidney transplant already have to use immunosuppressive drugs, and they are still at risk of recurrent diabetic kidney disease and other complications of diabetes. Islet transplantation in these patients has only rarely been successful in the past in part because the usual immunosuppressive drugs used in kidney transplantation cause diabetes and actually harm the transplant kidney in other ways. The immunosuppressive drugs used in the Edmonton Protocol are less likely to cause diabetes and are also less harmful to the kidney. In the second part of this project (Group 2), we will transplant islets into kidney transplant patients after they have switched to the immunosuppressive medications used in the Edmonton Protocol. Even if some of the patients do not get islet transplants or still need insulin shots after islet transplantation, we expect to see improvement in kidney function and blood glucose control.

DETAILED DESCRIPTION:
We anticipate that successful islet transplantation will establish a group of islet cell transplant patients who have normal blood sugars and do not need insulin injections. Some of this group will have received a kidney transplant as well. All these patients will be studied in great detail along with other investigators in our islet cell program to understand better the mechanisms of efficacy and side effects of islet transplant and these new immunosuppressive drugs.

ELIGIBILITY:
Inclusion Criteria:

Type 1 diabetes for > 5 years AND Hypoglycemia unawareness, not felt adequately by patient (glucose < 54mg/dL) in last 1.6 years, not otherwise explained, requiring outside help OR Metabolic lability/instability, characterized by hypoglycemia or ketoacidosis (>2 hospital < 12 mo), chaotic glucose profile (MAGE > 120mg/dL), disruption in lifestyle or danger to life, to self, to others OR Failure of intensive insulin management, as judged by an independent endocrinologist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States